CLINICAL TRIAL: NCT07345065
Title: The Sleep-MOMagement Project: Effectiveness of Person-centred Behavioural Interventions for Postpartum Maternal Sleep Improvement in Sleep-disturbed First-time Mothers.
Brief Title: Sleep-MOMagement: Improving Postpartum Sleep in First-time Mothers Through Tailored Behavioral Approaches.
Acronym: SleepMOM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: De deyne Manon (Other)
Collaborators: Vrije Universiteit Brussel (Other); KU Leuven (Other)
Responsible Party: Sponsor-Investigator, De deyne Manon, PhD researcher, Research Foundation - Flanders (Fonds Wetenschappelijk Onderzoek)
Organization: Research Foundation - Flanders (Fonds Wetenschappelijk Onderzoek) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FWOSB185
Record Dates: First submitted 2025-12-11; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Insomnia
Keywords: postpartum; sleep; insomnia; physiotherapy; behavioural; physical activity; women; circadian
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study protocol outlines a parallel group (1:1:1) randomized controlled trial with an embedded qualitative component.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment As Usual (No Intervention): The control group receives Treatment as Usual (TAU) based on standard postnatal care guidelines. As sleep management and physical activity are typically not part of these guidelines, this group serves as a 'waiting-list' control. After the study concludes, TAU participants are provided with BSM and BAET materials.
- BSM (Experimental group 1) (Experimental)
  Interventions: Behavioral: Behavioural Sleep Managament
- BAET (Experimental Group 2) (Experimental)
  Interventions: Behavioral: Behavioural Aerobic Exercise Therapy

INTERVENTIONS:
Behavioral: Behavioural Sleep Managament — The Behavioural Sleep Management intervention is provided by a master level physiotherapist and consists of sleep-focused psychoeducation, stimulus control, sleep hygiene, relaxation techniques, addressing unhelpful beliefs related to sleep , prioritizing self-care, checking for social support, and infant settling. The delivered form is based on CBT-I guidelines. Importantly, this intervention is not a form of psychotherapy. It does not involve exploration of emotional themes unrelated to sleep, diagnostic work, or cognitive restructuring beyond sleep-specific themes. Instead, it focuses on practical, educational, and behavioural strategies aimed at improving sleep quality and habits. Additionally, the intervention deliberately omits the time-in-bed restriction component typically found in standard CBT-I. This intervention is delivered through four appointments over a six-week period, supplemented with informational graphics and booklets that are sent via e-mail.
  Arms: BSM (Experimental group 1)
Behavioral: Behavioural Aerobic Exercise Therapy — The Behavioural Aerobic Exercise Therapy intervention is delivered by a master level physical therapist and primarily targets the daytime physical activity behaviour of the women. It includes coaching sessions focused on providing the necessary knowledge, skills, and support to implement an individually tailored aerobic exercise program and to adopt and sustain a physically active lifestyle. This intervention model aligns with the guidelines established by the American College of Sports Medicine. This intervention is delivered through four appointments over a six-week period, supplemented with informational graphics and booklets that are sent via e-mail.
  Arms: BAET (Experimental Group 2)

SUMMARY:
The goal of this clinical trial is to find out if person-centered behavioral interventions can help first-time mothers sleep better after childbirth. The study compares two approaches-a behavioral sleep management program and a behavioral aerobic exercise program-to usual postpartum care for women experiencing insomnia symptoms.

The main clinical outcome is insomnia severity. The study also evaluates economic outcomes, including healthcare use, work absenteeism, overall health utility.

Participants will:

* Receive one of the interventions or continue with usual care.
* Keep a sleep diary, a diary on physical activity, and complete questionnaires about sleep, mood, daily functioning, psychosocial factors, and economic outcomes.
* Follow the program instructions, which may include sleep strategies or guided aerobic training, depending on the group.

DETAILED DESCRIPTION:
* The primary objective of this study is to compare the clinical and cost-effectiveness of two behavioural interventions against treatment as usual (TAU) for postpartum women experiencing (sub)clinical insomnia. The study will assess insomnia severity as the primary clinical outcome and healthcare use as the primary economic outcome at six months post-intervention.
* Secondary objectives of this trial are: (1) To define clinical, therapeutic, and sociodemographic factors acting as predictors or moderators for treatment response on insomnia severity in postpartum women. (2) To assess baseline associations between insomnia symptoms, pain, symptoms of depression, and anxiety, and sleep outcomes. (3) To conduct a qualitative process evaluation to explore the experiences and perceptions of participants and intervention providers, as well as examining the underlying mechanisms and contextual factors that influence the effectiveness of the interventions under investigation.
* The primary endpoint was chosen at 6 months follow-up (T3). Other endpoints involve T0 (baseline data), T1 (immediate post-intervention data), and T2 (3 months follow up).
* A total of 135 postpartum women with (sub)clinical insomnia are recruited from community areas around Brussels and Leuven (Belgium) through a combination of community and internet-based strategies. Flyers are distributed across the University Hospitals of Brussels and Leuven, as well as in maternal and child health services, daycare centers, pharmacies, GP waiting rooms, and other key locations frequented by new mothers within a 30 km radius of these cities. Social media advertisements are also placed in relevant parent and perinatal groups. Interested women can contact the research team via phone, email, or a contact form.
* Participants are screened through a phone interview conducted by a researcher not involved in the randomization process. Screening is based on validated questionnaires described in the protocol. Eligible participants receive an informed consent form via email and are instructed to provide a signed copy before enrollment in the study.
* A total of 135 participants are randomized into three groups using block randomization by an independent researcher who is not involved in the trial delivery. To maintain balanced groups, participants are stratified by infant age and insomnia severity.
* Both experimental interventions are delivered by physiotherapists over a six-week period, supplemented with additional materials and a booster call at 3 months post-intervention. The control group receives Treatment as Usual (TAU). After the study concludes, TAU participants are provided with the intervention materials.
* To ensure the fidelity and quality of the delivered interventions, sessions will be audio- or video-recorded with participant permission. A random selection of recordings will be independently reviewed by two researchers using predefined criteria.
* Quantitative data will be collected via web-based self-reported questionnaires using REDCap at T0, T1, T2, and T3. Objective data on sleep and physical activity will also be gathered using wrist-worn actigraphy devices. Recruitment and follow-up require collection of participants' names and contact details. Demographic information is collected at T0.
* Data on therapy dose, adherence, and delivery will be collected through logbooks and recordings. Participants' perceptions of the interventions will be evaluated via surveys and open-ended questions at 3 and 6 months follow-up.
* Handling of missing data: Participants receive automated reminders and personal follow-ups. Appropriate imputation techniques will be used, with likelihood-based estimation assuming data are missing at random.
* Analyzing treatment effectiveness: The primary outcome (insomnia severity) will be analyzed using a linear mixed model. Analyses will follow an intention-to-treat approach. Results will be reported with mean differences, confidence intervals, p-values, and effect sizes.
* Longitudinal daily data will be analyzed with the Group Iterative Multiple Model Estimation (GIMME) approach to capture within- and between-person dynamics.
* Cost-effectiveness and cost-utility analyses will be conducted from a societal perspective, following KCE guidelines.
* Additional explorative analyses and post-hoc analyses will investigate predictors, moderators, and associations between outcomes.
* Process evaluation: Both qualitative and quantitative data will be analyzed to assess intervention fidelity, adherence, and participants' experiences. Findings will be integrated through triangulation to provide a comprehensive understanding of the interventions' impact.
* DATA MANAGEMENT: Data collection and storage will be overseen by the coordinating investigator under supervision of the principal investigators. All questionnaire data will be securely stored in REDCap. Pseudonymized data, logbooks, actigraphy data, and recordings will be stored on secured institutional servers.
* DATA STORAGE: After study completion, all data will be archived in the VUB Institutional Repository and the KU Leuven Research Data Repository for 25 years under restricted access.
* Personal identifiable information (PII) will be assigned unique IDs and stored separately from study data. Only the coordinating team will have access to the identification log. Data will only be shared in pseudonymized or aggregated form.
* Declaration of Helsinki: The trial will adhere to the Declaration of Helsinki, Good Clinical Practice, the protocol, and applicable laws.
* Ethics Committee: Approval of the protocol, informed consent forms, and other relevant documents will be obtained from the applicable ethical committees before the start of the trial.
* Informed Consent: Written informed consent must be provided by each participant prior to any study-related activities.
* Privacy: Data collection and processing will be limited to necessary information, with confidentiality safeguarded according to applicable laws. Participants will be identified only by study numbers in reports and sponsor communications.

ELIGIBILITY:
Inclusion Criteria:

Women are eligible for study participation if they:

* (1) Have had a singleton pregnancy.
* (2) Are between 4 to 12 months postpartum with their first child.
* (3) Exhibit (sub)clinical insomnia, operationalized as an Insomnia Severity Index (ISI) score greater than 7 7 and having answered 'yes' on the following three statements: a) I have trouble falling asleep, and/or staying asleep and/or I have early morning awakenings AND this causes daytime symptoms. b) My sleeping problem is not caused by an external factor (the baby or my partner). c) These sleeping problems occur at least 3 times a week for at least 3 months.
* (4) Have access to a telephone, computer, and email.
* (5) Possess adequate Dutch literacy to comprehend therapy content, questionnaires, and instructions.

Exclusion Criteria:

Women are excluded from participation if they:

* (1) Are currently pregnant.
* (2) Are shift workers.
* (3) Have severe diagnosed psychopathologies (e.g., bipolar disorder, post-traumatic stress disorder, psychosis)
* (4) Have current severe or untreated sleep disorders (narcolepsy, restless legs syndrome, circadian rhythm disorders)
* (5) Have an unstable medical condition that may disrupt sleep.
* (6) Have received cognitive-behavioural therapy for insomnia (CBTi) within the last 6 months.
* (7) Experience sleep deprivation due to unsettled infant sleep/wake behaviour, defined as the infant waking more than three times per night for more than 30 minutes and requiring parental support to re-initiate sleep.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity | This outcome will be measured at the following endpoints: - T0 = Day 0 - T1 = Day 42 - T2 = Day 132 - T3 = Day 222 The primary endpoint is the difference between T0 and T3.
  This outcome will be measured using the Insomnia Severity Index, a self-reporting questionnaire that evaluates the severity of insomnia symptoms over the past month through 7 items, each rated on a 0-4 scale. Higher total scores reflect greater insomnia severity.
Economic evaluations: Medical Consumption | This outcome will be measured at the following endpoints: - T0 = Day 0 - T3 = Day 222
  Medical Consumption Questionnaire (MCQ): A self-reporting generic (non-disease specific) questionnaire that identifies the direct costs of medical care, consisting of 29 questions.
Economic evaluations: Productivity Cost | This outcome will be measured at the following endpoints: - T0 = Day 0 - T3 = Day 222
  Productivity Cost Questionnaire (PCQ): A self-reporting questionnaire consisting of 3 aspects 1) absenteeism, 2) presenteeism, and 3) productivity losses associated with unpaid work.
Economic evaluations: Health-related quality of life | This outcome will be measured at the following endpoints: - T0 = Day 0 - T3 = Day 222
  EQ-5D-5L: A self-reporting questionnaire for measuring health-related quality of life, consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and 5 levels (no problems, slight problems, moderate problems, severe problems, extreme problems).

SECONDARY OUTCOMES:
Sleep Quality | This outcome will be measured at the following endpoints: T0 = Day 0 T1 = Day 42 T2 = Day 132 T3 = Day 222
  This outcome will be measured using the Pittsburgh Sleep Quality Index (PSQI), a self-reporting questionnaire that evaluates sleep quality over the past month, consisting of 7 subscales: subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medication, daytime dysfunction. The individual scores for the 7 subscales are ultimately summed to obtain a total PSQI score (ranging from 0 to 21). A higher total score indicates poorer sleep quality.
Sleep Propensity | This outcome will be measured at the following endpoints: T0 = Day 0 T1 = Day 42 T2 = Day 132 T3 = Day 222
  This outcome will be measured using the Epworth Sleepiness Scale (ESS), a self-reporting questionnaire, consisting of 8 items that describe specific situations in which individuals rate their likelihood of dozing off or falling asleep. Each situation is scored on a scale from 0 (no chance of dozing) to 3 (high chance of dozing), with higher total scores indicating greater daytime sleepiness.
Fatigue | This outcome will be measured at the following endpoints: T0 = Day 0 T1 = Day 42 T2 = Day 132 T3 = Day 222
  This outcome will be measured using the Brugmann Fatigue Scale (BFS), a self-reporting questionnaire that evaluates mental and physical fatigue and focuses specifically on rest propensity. It consists of 8 items, each scored on a 4 point Likert scale with higher scores indicating more severe fatigue.
Sleep-related beliefs and attitudes | This outcome will be measured at the following endpoints: T0 = Day 0 T1 = Day 42 T2 = Day 132 T3 = Day 222
  Dysfunctional Beliefs and Attitudes about Sleep Scale - 16 (DBAS-16), a self-reporting 16-item questionnaire designed to assess unhelpful or disruptive beliefs and attitudes about sleep that can contribute to insomnia. It uses a simple Likert-type response scale (0-10).
Chronotype | This outcome will be measured at the following endpoints: T0 = Day 0 T2 = Day 132 T3 = Day 222
  Oginska Chronotype Questionnaire, a questionnaire designed to assess an individual's chronotype, which reflects their natural preference for sleep and activity timing. It classifies individuals into morning types, evening types, or intermediate types, providing insight into their circadian rhythm and its influence on daily functioning, mood, and performance.
Circadian alignment of food intake | This outcome will be measured at the following endpoints: T0 = Day 0 T2 = Day 132 T3 = Day 222
  Chrononutrition Profile Questionnaire: A self-reporting tool designed to evaluate an individual's eating patterns in relation to their circadian rhythms. It assesses factors such as meal timing, frequency, and consistency.
Pain severity and interference | This outcome will be measured at the following endpoints: - T0 = Day 0 - T1 = Day 42 - T2 = Day 132 - T3 = Day 222
  Brief Pain Inventory (BPI): A self-reporting questionnaire that assesses pain severity and its impact on daily functioning. It comprises two main sections: pain intensity and pain interference, with each item rated on a scale from 0 to 10, where higher scores indicate greater pain.
  In this study, we use a modified version in which the time frame is set to one month, ensuring the questionnaire specifically captures average pain experiences over the past four weeks, as well as at the time of assessment. Additionally, extra questions have been included to assess the nature of the pain, allowing respondents to indicate whether their pain is chronically present or occurs in recurrent episodes.
Depressive symptoms | This outcome will be measured at the following endpoints: - T0 = Day 0 - T1 = Day 42 - T2 = Day 132 - T3 = Day 222
  Edinburgh Postnatal Depression Scale (EPDS): A self-reporting questionnaire that assesses symptoms of postnatal depression. The questionnaire consists of 10 items, asking mothers about their mood and feelings over the past month (adapted time frame). Each item is scored from 0 to 3, with higher scores indicating a greater risk of postnatal depression.
Anxiety | This outcome will be measured at the following endpoints: - T0 = Day 0 - T1 = Day 42 - T2 = Day 132 - T3 = Day 222
  Generalized Anxiety Disorder scale - 7 (GAD-7): A brief, seven-item questionnaire used to screen for and assess the severity of generalized anxiety disorder (GAD). Scores range from 0 to 21, with higher scores indicating more severe anxiety.
Physical Activity | This outcome will be measured at the following endpoints: - T0 = Day 0 - T1 = Day 42 - T2 = Day 132 - T3 = Day 222
  International Physical Activity Questionnaire Short-Form (IPAQ-SF): A self-reporting questionnaire that assesses the intensity, type, and level of physical activity over the past month (adapted time-frame from the original questionnaire). It consists of 7 short questions.
Maternal Quality Of Life | This outcome will be measured at the following endpoints: - T0 = Day 0 - T2 = Day 132 - T3 = Day 222
  Maternal Quality of Life Instrument (MPQoL-I): A self-reporting questionnaire that assesses the satisfaction of mothers with their postpartum life, consisting of 16 items.
Expectancy of treatment | This outcome will be measured at the following endpoints: - T0 = Day 0 - T1 = Day 42 - T3 = Day 222
  Credibility Expectancy Questionnaire (CEQ): A self-reporting, brief questionnaire measuring cognitive credibility and affective expectancy, consisting of 6 questions, widely used in clinical trials.
Therapeutic Working Alliance | This outcome will be measured at the following endpoints: - T0 = Day 0 - T1 = Day 42 - T3 = Day 222
  Working Alliance Inventory (WAI): A self-reporting questionnaire that evaluates the therapeutic alliance both from a within-person and a between-person perspective. It consists of 36 items.
Self-efficacy | This outcome will be measured at the following endpoints: - T0 = Day 0 - T1 = Day 42 - T3 = Day 222
  General Self-Efficacy Scale (GSES): A self-reporting questionnaire measures an individual's belief in their ability to manage stress and challenging situations, consisting of 10 items. Each item is scored on a 4-point Likert scale, with higher total scores reflecting greater self-efficacy.
Objective sleep parameters | Participants will wear the actigraph during 1 week at baseline, after the intervention period, at 3 months followup and at 6 months followup.
  Actigraphy (wrist-worn) measures sleep duration, sleep onset latency, wake after sleep onset (WASO), sleep efficiency, number of awakenings, and circadian rhythm metrics.
Objective physical activity parameters | Participants will wear the actigraph during 1 week at baseline, after the intervention period, at 3 months followup and at 6 months followup.
  Actigraphy (wrist-worn) measures total daily activity counts, time spent in activity intensity zones, sedentary time, daily energy expenditure estimates (METS/min)

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Vrije Universiteit Brussel, Health Campus, Department of Physiotherapy, Brussels, Jette
  - KU Leuven, Departement of Physiotherapy, Leuven, Leuven

IPD SHARING:
Plan to Share IPD: Undecided